CLINICAL TRIAL: NCT06330935
Title: Clinical Trial Evaluating the Effect of Tranexamic Acid on the Clinical Outcomes in Pediatric Patients With Traumatic Brain Injury
Brief Title: Evaluating the Effect of Tranexamic Acid on the Clinical Outcomes in Patients With Traumatic Brain Injury
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Lecturer of Clinical Pharmacy- Faculty of Pharmacy - Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 192-2023
Record Dates: First submitted 2024-02-18; First posted 2024-03-26 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TXA dose A arm (Active Comparator): Subjects will receive a 15 mg/kg bolus of Tranexamic acid over 20 minutes followed by 2 mg/kg/hr. infusion over 8 hours. The maximum bolus dose is 1000 mg, the maximum rate of infusion is 50 mg/min, and the maximum total maintenance dose is 1000 mg
  Interventions: Drug: Tranexamic Acid (TXA)
- TXA dose B arm (Active Comparator): Subjects will receive a 30 mg/kg bolus of Tranexamic acid over 20 minutes followed by 4 mg/kg/hr. infusion over 8 hours. The maximum bolus dose is 2000 mg, the maximum rate of infusion is 100 mg/min, and the maximum total maintenance dose is 2000 mg
  Interventions: Drug: Tranexamic Acid (TXA)
- Placebo arm C (Placebo Comparator): Subjects in the placebo group will receive a bolus dose of normal saline over 20 minutes followed by a normal saline infusion over 8 hours (in the same weight-based volume as the other study arms)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — 30 patients will be randomized to A arm and 30 patients to B arm
  Other Names: TXA dose A arm &TXA dose B arm
  Arms: TXA dose A arm; TXA dose B arm
Drug: Normal saline — 30 patients will be randomized this arm C
  Other Names: Placebo arm C
  Arms: Placebo arm C

SUMMARY:
Evaluate the effect of tranexamic acid on mortality in pediatric patients with traumatic brain injury. This could potentially lead to improved treatment protocols and better outcomes for this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

1. Age Less than 18 years old
2. Clinical diagnose of trauma to the Head and GCS score less than or equal to 13 with associated intracranial haemorrhage on cranial CT scan
3. Time of admission within 3 hour of injury.

Exclusion Criteria:

1. Patient Known pregnancy.
2. patient had Cardiac arrest prior to randomization
3. GCS score of 3 with bilateral unresponsive pupils
4. Known bleeding/clotting disorders.
5. Known seizure disorders.
6. Known history of severe renal impairment
7. Unknown time of injury
8. Prior TXA for current injury
9. Known venous or arterial thrombosis

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
The early traumatic brain injury-related death in the hospital | 24 hour and 48 hour after injury
  2. Decreasing the rate of early head injury-related death (within 24 hour after injury)
The difference between treatment group in the Intracranial haemorrhage growth | 24 hour
  We will measure intracranial hemorrhage progression at 24 hours in all subjects with intracranial hemorrhage on the initial clinical CT scan
The difference between the treatment groups in the incidence of mortality | 28 days
  Decreasing the rate of head injury-related death in hospital within 28 days of injury all-cause and cause-specific mortality, disability, vascular occlusive events (myocardial infarction, stroke, deep vein thrombosis, and pulmonary embolism)

SECONDARY OUTCOMES:
Need for neurosurgical management | 28 day
  Evacuation of acute subdural hematoma,Evacuation of epidural hematoma and Evacuation of traumatic intracerebral hematoma (contusions)
Days in the intensive care unit | 28 day
  Decreasing days in intensive care unit within 28 day of injury
Need for blood transfusion | 48 hour
  Decreasing the total amount of blood products transfused in the initial 48 hours following randomization. Blood product transfusion volume will be measured at 24 hours, 48 hours. This will include volume of packed red blood cells, plasma, platelets, and cryoprecipitate in mL/kg.
Adverse events | 28 days
  Decreasing incidence of seizures, complications and other adverse events
Pediatric Quality of Life (PedsQL) | 6 months
  Improving the Paediatric Quality of Life (PedsQL) . The PedsQL is a continuous score that ranges from 0-100.
Pediatric Glasgow Outcome Scale Extended (GOS-E) Peds) | 6 months
  Improving the Pediatric Glasgow Outcome Scale Extended (GOS-E Peds) scores

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University Hospital in New Damietta, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No